# Clinical Trial to Evaluate ET-01 in Subjects with Lateral Canthal Lines

Protocol No.: ET-01-LCL-206

incl. Amendment 2 NCT03326856

Apr. 23, 2018

Eirion Therapeutics, Inc. 25-K Olympia Ave., Suite 200 Woburn, MA 01801

Tel: 215-356-7532 Fax: 888-664-2736

The confidential and proprietary information in this document is provided to you as a Principal Investigator or consultant for review by you, your staff, and the applicable Institutional Review Board/Independent Ethics Committee or duly authorized representatives of the U.S. Food and Drug Administration under the condition that they are requested to keep it confidential. Your acceptance of this document constitutes agreement that you will not disclose the information contained herein to others without authorization from the Sponsor, Eirion Therapeutics, Inc.

# **TABLE OF CONTENTS**

| A | BBREVI | ATIONS | 5 |
|---|---|---|---|
| 1 | INTR | ODUCTION AND BACKGROUND | 6 |
| 2 | STU | DY OBJECTIVES AND PURPOSE | 7 |
| 3 | STU | DY DESIGN | 7 |
| | 3.1 | Overall Design | 7 |
| | 3.2 | Treatment Groups / Sample Size | 7 |
| | 3.3 | Efficacy Parameters and Timing | 7 |
| | 3.4.1<br>3.4.2<br>3.4.3<br>3.4.4<br>3.4.5<br>3.4.6<br>3.4.7<br>3.4.8 | Muscle Weakness or Paralysis Hematology Clinical Chemistry ECG Testing Immunogenicity Photography Treatment Procedure | 8<br>8<br>8<br>9<br>9 |
| | 3.5 | Study Visits and Procedures | 10 |
| | 3.6 | Measures to Minimize/Avoid Bias | 10 |
| 4 | MED | ICATION AND DOSING | 11 |
| | 4.1 | Dose Rationale | 11 |
| | 4.2 | Treatment of Subjects | 11 |
| | 4.3<br>4.3.1<br>4.3.2 | 99 | 14 |
| 5 | SELI | ECTION AND WITHDRAWAL OF STUDY SUBJECTS | 15 |
| | 5.1 | Inclusion Criteria | 15 |
| | 5.2 | Exclusion Criteria | 15 |
| | 5.3 | Concomitant Medication | 16 |
| | 5.4 | Subject Withdrawal or Removal From Study | |
| | 5.4.1 | Subject Unblinding Procedures | 17 |
| 6 | STU | DY PROCEDURES | 17 |
| | 6.1.1<br>6.1.2<br>6.1.3<br>6.1.4 | Week 1 Visit (+/- 2 days) | 19<br>19 |
| | <b>₹</b> 1117 | | |

| | 6.1.5 | | |
|----------|-------|-----------------------------------------|----------|
| | 6.1.6 | 6 Week 12 Visit (+/- 7 days) | 21 |
| | 6.1.7 | Week 18 Visit (+/- 7 days) | 21 |
| | 6.1.8 | B Week 26 Visit (+/- 7 days) | 21 |
| | 6.1.9 | Study Exit / Early Termination | 22 |
| | 6.1.1 | 0 Unscheduled Visits | 22 |
| 7 | STU | DY DURATION AND CONDUCT | 22 |
| | 7.1 | Conduct of Study | 22 |
| | 7.2 | Duration of Study | 23 |
| | 7.3 | Stopping Rules | 23 |
| | 7.4 | Monitoring for subject compliance | 23 |
| 8 | ADV | ERSE EVENT REPORTING | 23 |
| | 8.1 | Definitions | |
| | 8.1.1 | · | |
| | 8.1.2 | · | |
| | 8.1.3 | | |
| | 8.1.4 | , | |
| | 8.2 | Adverse Event Follow-up | |
| | 8.2.1 | Pregnancy | 27 |
| 9 | STA | TISTICAL PLAN | |
| | 9.1 | Statistical Methods | |
| | 9.1.1 | <b>y</b> | |
| | 9.1.2 | . , , | |
| | 9.1.3 | | |
| | 9.1.4 | • | |
| | 9.2 | Subject Population(s) for Analysis | |
| | 9.2.1 | | |
| | 9.2.2 | | |
| | 9.3 | Significance | |
| | 9.4 | Termination Criteria | |
| | 9.5 | Deviation Reporting | 30 |
| 10 | DIRE | | |
| | | ECT ACCESS TO SOURCE DATA/DOCUMENTATION | 31 |
| 11 | QUA | LITY CONTROL AND QUALITY ASSURANCE | |
| 11<br>12 | | | 31 |
| | ETH | LITY CONTROL AND QUALITY ASSURANCE | 31<br>31 |

| 15 | INVESTIGATOR'S AGREEMENT | 34 |
|-----|-------------------------------------------|----|
| 16 | REFERENCES | 35 |
| APF | PENDIX A: CROW'S FEET WRINKLE SCALE | 36 |
| APF | PENDIX B: SIGNS OF BOTULINUM TOXIN SPREAD | 38 |
| APF | PENDIX C: PROCEDURE FOR COLOR PHOTOGRAPHY | 39 |
| APF | PENDIX D: IRRITATION SCORING | 40 |

#### **ABBREVIATIONS**

AE Adverse Event

ANCOVA Analysis of Covariance

ANOVA Analysis Of Variance

BoNTA Botulinum toxin, Type A

CFW Crow's Feet Wrinkle (scale)

eCRF Case Report Form

ECG Electrocardiogram

FDA Food and Drug Administration

GCP Good Clinical Practice

ICH International Conference on Harmonization

IGA Investigator's Global Assessment score

IRB Institutional Review Board

ITT Intent-to-Treat

IUD Intra-Uterine Device

LCL Lateral Canthal Lines

LOCF Last Observation Carried Forward

PP Per-Protocol

SAE Serious Adverse Event

SSA Subject Self-Assessment

#### 1 INTRODUCTION AND BACKGROUND

Over time, the actions of the facial musculature, coupled with loss of skin elasticity and a reduction in subcutaneous tissue, result in the development of facial lines. With the decrease in skin elasticity, repeated facial expressions can become permanent lines<sup>1</sup>. The periorbital area is one of the first places on the face to show signs of aging, in the form of lateral canthal lines or Crow's Feet. Genetic differences and environmental toxins, predominantly ultraviolet light exposure and cigarette smoking, may alter the rate of this normal aging process<sup>2</sup>.

Over the past two decades, there has been increasing demand for aesthetic procedures to reverse the effects of aging, particularly in the facial area, and treatment of Crow's Feet is among the most frequent of corrective treatment requests. A number of techniques have been developed to meet the increasing demand for aesthetic procedures to reverse the signs of aging. These include: incisional and excisional surgery, various resurfacing procedures, and the use of temporary or semi-permanent, injectable dermal fillers such as allogeneic or xenogeneic collagen, hyaluronic acid, and autologous fat cells. Topical agents, such as retinoic acids, glycolic acids and lactic acids, are other common methods to minimize Crow's Feet and other facial wrinkles.

Injection of *botulinum* toxin type A (BoNTA) is now one of the most common aesthetic procedures performed and there is a considerable body of medical literature demonstrating its safety and efficacy in aesthetic indications<sup>3</sup>. On a molecular level, *botulinum* toxin prevents the release of preformed mediators, such as acetylcholine, from motor nerve endings leading to a flaccid paralysis.

BoNTA is an effective treatment for Crow's Feet and is associated with high subject satisfaction. However, the treatment requires multiple injections into a well innervated, sensitive area that is prone to bleeding and bruising and close to delicate organs such as the eyes and lachrymal glands. In addition, misplacement of injection can lead to unwanted effects in non-target areas. Therefore, a topical dermatological formulation to deliver the active ingredient, avoiding the discomforts and potential side effects of injections, would be highly desirable.

Several studies have been conducted assessing the dose-response of the topical *botulinum* product, ET-01<sup>4</sup>, in the treatment of Crow's Feet. The product was well tolerated. This current clinical trial seeks to expand on the existing work.

Confidential

<sup>&</sup>lt;sup>1</sup> Ascher, B et al. Dermatol Surg 35:1478-1486, 2009

<sup>&</sup>lt;sup>2</sup> Carruthers, A et. al. Dermatol Surg 2008; 34:S173–S178

<sup>&</sup>lt;sup>3</sup> Coté, T. et al. J. Am. Acad. Dermatol. 2005;53:407-15

<sup>&</sup>lt;sup>4</sup> ET-01 was previously studied under Anterios' code ANT-1207 and ANT-1401

#### 2 STUDY OBJECTIVES AND PURPOSE

The purpose of this Phase 2 study is to provide evidence of the safety, tolerance, and efficacy of ET-01 in the treatment of lateral canthal lines (Crow's Feet).

Apr. 23, 2018

#### 3 STUDY DESIGN

## 3.1 Overall Design

The study will be an out-patient, prospectively randomized, double-blind, vehicle-controlled, dose-ranging clinical trial involving up to two centers. The study is planned as a sequential dose escalation trial. Each cohort will be fully enrolled and complete the Week 2 visit to allow for a safety review before initiating enrollment of the next dose group.

## 3.2 Treatment Groups / Sample Size

The following dose groups and sample sizes are planned:

| | | | ET- | 01 | | | Veh | icle | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Cohort | Dose | Dose | Precondition | | _ | Precondition | | | _ | N / | |
| | [units] | [ng] | Α | В | С | ۷ | Α | В | С | ۷ | cohort |
| 1 | 325 U | 1.2 | 3 | 3 | 3 | 9 | 1 | 1 | 1 | 3 | 12 |
| 2 | 585 U | 2.1 | 3 | 3 | 3 | 9 | 1 | 1 | 1 | 3 | 12 |
| 3 | 825 U | 3.0 | 3 | 3 | 3 | 9 | 1 | 1 | 1 | 3 | 12 |
| 4 | 1,150 U | 4.0 | - | 8 | - | 8 | - | 4 | - | 4 | 12 |
| Total | Σ = | | 9 | 17 | 9 | 35 | 3 | 7 | 3 | 13 | 48 |

A=AdminStamp 600, B=AdminStamp 900, C=AdminStamp 1,500

In Cohorts 1-3, the treatment area will be preconditioned with one of three AdminStamps, i.e. AdminStamp 600, 900, or 1500, according to the table above. In Cohort 4, the treatment area will be preconditioned with AdminStamp 900 only. ET-01 will be applied immediately after pre-conditioning.

# 3.3 Efficacy Parameters and Timing

Efficacy will be assessed using the Crow's Feet Wrinkle Scale (CFW), which is a published validated, photo-numeric guide that grades severity of lateral canthal lines into one of the five categories of 0=none, 1=minimal, 2=mild, 3=moderate, and 4=severe. (see Appendix A for details). Using the same scale, assessments will be made by both, the investigator (IGA) and the subjects (SSA). Assessments are made "static" to avoid recall bias.


The IGA is recorded separately for the right and left canthal areas, both "at rest" and "on contraction". The IGA will be recorded at each visit. The subject's self-assessment of the CFW score will also be recorded "at rest" and "on contraction" at each visit.

## 3.4 Safety Parameters and Timing

Safety will be assessed during the study by collection of study events, review of concomitant treatments and laboratory data. Clinical adverse event reporting will be conducted at each visit.

All laboratory measurements will be performed by a central laboratory using appropriate and validated methods. Values will be reported to the Investigator and the Sponsor. Laboratory reference range values will be described in the laboratory manual. Investigators will assess all out of range values as being clinically significant or not.

## 3.4.1 Vital signs

Weight, height (Screening visit only) temperature, resting pulse, blood pressure, and respiration rate. Vital signs will be recorded at every visit.

## 3.4.2 Muscle Weakness or Paralysis

Participants will be monitored for potential signs of *botulinum* induced muscle weakness or paralysis. Subjects will be evaluated for Signs of Botulinum Toxin Spread (muscle weakness - ocular and the extremities) or difficulty swallowing or breathing (cranial nerve assessment, Appendix B).

The neurologic assessments are made at Baseline, Week 1, Week 2 and Week 4.

#### 3.4.3 Hematology

Non-fasting clinical hematology evaluations are:

hemoglobin, hematocrit, red blood cell count, white blood cell count, with a differential, and a platelet count.

Non-fasting clinical hematology evaluations will be performed at Week 0 (Baseline), Week 4, and Week 26/End of Study.

## 3.4.4 Clinical Chemistry

A standard non-fasting chemistry panel will be performed which will include the following parameters:

glucose, uric acid, calcium, sodium, potassium, phosphorus, chloride, alkaline phosphatase, aspartate aminotransferase, alanine aminotransferase, total bilirubin,

bicarbonate, creatinine, blood urea nitrogen, lactate dehydrogenase, total protein, albumin.

The chemistry panel will be performed at Baseline (Week 0), Week 4, and Week 26/End of Study. A urine pregnancy test will be performed for women of child-bearing potential at Baseline and the Week 4 visit.

## 3.4.5 ECG Testing

A 12-lead ECG will be recorded measuring the RR, PR, QRS, and QT interval durations prior to treatment application at Baseline and at Week 2.

## 3.4.6 Immunogenicity

Plasma samples will be banked for future analysis of anti-botulinum serum antibodies as a safety parameter for possible immunization against botulinum.

Samples will be taken at Baseline, Week 4, and Week 26.

## 3.4.7 Photography

Color photographs will be taken at every visit. Five pictures will be taken as described in Appendix C.

#### 3.4.8 Treatment Procedure

To capture the level of comfort or discomfort caused by the skin pre-treatment with the AdminStamps and subsequent rubbing in of the study medication subjects will be asked to rate their experience on a scale from "-5" (very bad) to "+5" (very good).



## 3.5 Study Visits and Procedures

A schematic study diagram is shown below:

| Procedure | Scr./BL | W 1 | W 2 | W 4 | W 8 | W 12 | W 18 | W 26 | |
|---|---|---|---|---|---|---|---|---|---|
| | Day 0<br>± 0 | Day 7<br>± 2 | Day<br>14<br>± 3 | Day<br>28<br>± 4 | Day<br>56<br>± 7 | Day<br>84<br>± 7 | Day<br>126<br>± 7 | Day<br>182<br>± 7 | End of<br>Study# |
| Informed Consent | Х | | | | | | | | |
| Assess Eligibility & Medical History | Х | | | | | | | | |
| Review Con-meds | Х | Х | Х | Х | Х | Х | Х | Х | |
| Record AEs | Х | Χ | Х | Х | Х | Х | X | Х | |
| Weight and Vital<br>Signs | Х | Х | X | Х | Х | Х | Х | Х | |
| Signs of Botulinum<br>Spread | Х | Х | Х | Х | | | | | |
| Hematology and Chemistry | Х | | | Х | | | | | Х |
| Anti-Botulinum<br>Antibodies | Х | | | Х | | | | | Х |
| Urine Pregnancy test (WOCBP) | Х | | | Х | | | | | |
| ECG | Х | | Х | | | | | | |
| IGA Score | Х | Х | Х | Х | Х | Х | Х | Х | |
| Subject Self-<br>Assessment (SSA) | Х | Х | X | Х | Х | Х | Х | Х | |
| Photography | Х | Х | Х | Х | Х | Х | Х | Х | |
| Randomization | Х | | | | | | | | |
| Apply Study<br>Medication | Х | | | | | | | | |

<sup>#</sup> also for early termination

The study will consist of up to 8 office visits.

## 3.6 Measures to Minimize/Avoid Bias

To minimize bias, subjects will be randomly allocated to one of the two treatment groups, i.e. active vs. vehicle, within each dosing cohort. Neither subjects nor investigators will be aware of the treatment allocation. Pre-treatment will also be randomly allocated.

Preparation of study medication, skin pre-conditioning, and drug application will be done by a person different from the investigator making the wrinkle assessments.

#### 4 MEDICATION AND DOSING

#### 4.1 Dose Rationale

Finding evidence of a safe and effective dose is the purpose of this study. In previous clinical studies doses of up to 7.4 ng (2,000 U) were applied under occlusion and were well tolerated. Likewise, in another study ET-01-SPC-101, that is still ongoing, using the same AdminStamp micro-needle arrays for skin pre-conditioning, no safety concerns other than temporary low grade redness/irritation have emerged. The current study continues to explore the dose-response relationship conservatively escalating doses at factor 1.4.

## 4.2 Treatment of Subjects

The study preparation or vehicle consists of a milky, white lotion of low viscosity. The drug product and diluents will be provided in kits containing identical 3 mL dropper bottles that contain 1.0 mL of either ET-01 at the appropriate concentration or Vehicle.

The following dose groups and sample sizes are planned:

| | | | ET- | 01 | | | Veh | icle | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Cohort | Dose | Dose | Precondition | | Precondition _ Precondition _ | | Precondition | | | _ | N/ |
| | [units] | [ng] | Α | В | С | ۷ | Α | В | С | ۷ | cohort |
| 1 | 325 U | 1.2 | 3 | 3 | 3 | 9 | 1 | 1 | 1 | 3 | 12 |
| 2 | 585 U | 2.1 | 3 | 3 | 3 | 9 | 1 | 1 | 1 | 3 | 12 |
| 3 | 825 U | 3.0 | 3 | 3 | 3 | 9 | 1 | 1 | 1 | 3 | 12 |
| 4 | 1,150 U | 4.0 | - | 8 | - | 8 | - | 4 | - | 4 | 12 |
| Total | Σ = | | 9 | 17 | 9 | 35 | 3 | 7 | 3 | 13 | 48 |

A=AdminStamp 600, B=AdminStamp 900, C=AdminStamp 1,500

Randomization to a treatment group within each cohort will be obtained following a randomization list prepared by the Sponsor. Likewise, randomization to a pre-treatment, i.e. type of Admin Stamp will be obtained following a randomization list prepared by the Sponsor.

The study medication will be applied TOPICALLY and only to subject's canthal areas. Before study medication is brought into the treatment room, make sure that no syringes or needles are present.

The treatment area is the periorbital region in the distribution of the muscles responsible for the Crow's Feet wrinkles. The muscle being treated to reduce the Crow's Feet wrinkle – the *orbicularis oculi* – is illustrated Figure 1.

Figure 1: M. orbicularis oculi



In general, the treatment region begins on the bony rim of the orbit, extending laterally to approximately one centimeter from the exterior edge of the hairline, 1 - 1.5 cm above and 1.5 - 2 cm below a horizontal line emanating from the lateral canthus to the hairline. This area of application is illustrated by the black outline in the picture below:

Figure 2: Treatment Area



As a guide to treatment, it is helpful to have the subject contract the orbicularis oculi muscle by asking the subject to produce a maximal smile so that the muscular extension can be visualized for that subject's treatment. In no case, however, should ET-01 ever be applied within the area circumscribed by the interior edge of the orbital rim.

The treatment area will be pre-conditioned by pressing the AdminStamp <u>firmly</u>, applying approximately 3-4 pounds of pressure, to the skin. The location of the areas of pre-conditioning are illustrated by the blue circles in Figure 2. There will be five (5) overlapping impressions made along the bony rim of the orbital cavity and two (2) impressions distal and inferior to the horizontal mid-line. After all seven impressions have been made, the micro-needle array will be rotated by approximately 90° and the process is repeated.

Immediately thereafter, using a gloved finger, the investigator will massage the topical treatment into the skin of the treatment area.

The medication is of low viscosity and administered one drop at a time to avoid run-off. As an additional precaution, the subject will be positioned on an examination table or fully reclined examination chair such that his/her temple will slightly slant backwards and to the side, directing any run-off away from the eyes and into the hairline. The subject will be instructed to close his/her eyes which will then be covered with eye covers, e.g., IPL-Aid™ Disposable Eye Shields, and an absorbent paper or cloth. The clinical investigator will wipe the periorbital region with an alcohol wipe and then dry thoroughly with a cotton swab.

There are 3 phases that the study drug will go through before it is completely absorbed into the skin. The clinical investigator will be instructed to make sure to visually observe all 3 phases during application process before additional small aliquots of Test Article are applied as listed below:

Phase 1: Gelling the sample becomes clear in color and flowable.

Phase 2: Creaming the sample becomes more viscous, is white in color, and

sticky.

Phase 3: Absorption the sample becomes clear in color and has a glossy smooth

finish. There is no visible residue left on the skin after

absorption.

The process of treatment application will take approximately 5 -10 minutes each. This procedure will be completed when there is no liquid visible on the surface of the skin.


This procedure will be employed for both, the right and left periorbital regions. The start and finish time will be recorded in the eCRF. The study medication kit drug label will be completed and peeled-off for application in the subject's Case Report Form.

## 4.3 Drug Storage and Drug Accountability

## 4.3.1 Drug Storage

The investigator will ensure that the investigational product is stored in appropriate conditions in a secure, locked refrigerator with controlled access. Until ready for dispensing, the investigational product will be stored at a controlled temperature of +5°C. Temperature logs will be maintained to document that the storage temperature has not deviated from the recommended range. Should a deviation occur in the storage temperature of unopened investigational product kits, the investigator will complete and submit an Investigational Product Deviation Report form by e-mail or fax to the Sponsor. The Sponsor will review the information submitted and will provide direction regarding further use of the applicable kit/s.

## 4.3.2 Drug Accountability

The principal investigator at each site is responsible for maintaining accurate records of the receipt and application of all investigational materials. The investigator may apply the investigational drug only to eligible subjects enrolled in the study. All applications of the investigational drug will be conducted at the study sites.

Eirion Therapeutics will provide drug accountability forms to assist the investigator in maintaining current and accurate inventory records covering receipt, application, and the return of investigational drug supplies. When a shipment is received, the investigator or designee will verify the quantities received. The Case Report Form includes the identification of the person to whom the drug is applied, the date of application, and any returned or unused drug. These records will be readily available for inspection by the Sponsor or a monitor and are open to any other regulatory authority inspection at any time.

When the supplies are returned, the investigator, designee, or monitor signs the investigational drug return log to verify that all used, unused, or partially used supplies have been returned, and that no study supplies remain in the investigator's possession. One copy of all inventory records and the return statement are retained by the investigator for the study files.

At study termination, unless otherwise specified, all used, unused, and partially used drug supplies should be returned to the distribution center. The study drug return form will be returned to Eirion Therapeutics, Inc., and a copy will be maintained on site.

#### 5 SELECTION AND WITHDRAWAL OF STUDY SUBJECTS

The study will enroll adult male and female subjects diagnosed with mild to severe Crow's Feet.

#### 5.1 Inclusion Criteria

- able to understand and give written informed consent
- 25 65 years of age
- willing to have facial pictures taken per protocol
- minimal to moderate Crow's Feet wrinkles (IGA 1-3) at rest
- moderate to severe Crow's Feet (IGA 3-4) on contraction
- moderate to severe Crow's Feet (SSA 3-4) on contraction
- Have adequate vision without the use of eyeglasses to assess facial wrinkles in a mirror (contact lenses are OK)
- willingness to refrain from the use of facial fillers, retinoids, Botox, laser treatments, or any product affecting skin remodeling or that might cause an active dermal response during the course of the study
- female subjects must have a negative urine pregnancy test and be non-lactating at the Baseline visit
- female subjects must utilize one of the following methods of birth control
  throughout the study: IUD, diaphragm, a condom, a spermicidal gel or foam, oral
  contraceptives (provided subject has been utilizing this method for at least
  3 months prior to baseline and has not changed the brand within this period), or
  patch, injectable, implantable, or vaginal ring contraceptives. Subjects may also
  participate if they are surgically sterilized (tubal sterilization or hysterectomy).
- subjects should be in good general health as determined by the investigator and free of any disease that may interfere with study evaluations or the Investigational Product

#### 5.2 Exclusion Criteria

- history of adverse reactions to any prior botulinum toxin treatments
- history of vaccination with botulinum toxin
- history of non-response to any prior botulinum toxin treatments
- botulinum toxin treatment in the prior 6 months
- history of periocular surgery, brow lift or related procedures

- soft tissue augmentation or any procedures affecting the lateral canthal region in the prior 12 months
- dermabrasion or laser treatment in the periocular region in the last 6 months
- topical prescription-strength retinoids in the prior 3 months to the treatment area
- application of any topical prescription medication to the treatment area within 14 days prior to treatment
- subjects on clinically significant, concomitant drug therapy (See section 5.3 below).
- present or history of neuromuscular disease, eyelid ptosis, muscle weakness or paralysis
- present or history of "dry eye"
- systemic aminoglycoside use in the week prior to treatment application
- participation in another investigational drug trial or receiving any investigational treatment(s) within 30 days of Baseline
- alcohol or drug abuse within the past 3 years
- female subjects who are pregnant or are nursing a child
- psychiatric disease interfering with the subject's ability to give informed consent
- refusal or inability to comply with the requirements of the protocol for any reason

#### 5.3 Concomitant Medication

Any prescription or over-the-counter medication taken during the study will be recorded in the appropriate section of the Case Report Form.

The following medications are prohibited:

- Botulinum toxin containing products for the course of the study
- The use of any facial fillers, laser treatments, or any product affecting skin remodeling for the course of the study
- Dermabrasion or laser treatment in the periocular region for the course of the study
- Topical prescription-strength retinoids in the periocular region for the course of the study
- Tanning booths or sun exposure for the treatment day and the following 2 days
- Any topical medications applied to the treatment area for the day of treatment and 5 days following treatment. Toiletry and make-up are permitted.
- Systemic aminoglycosides for the day of treatment and 7 days following the treatment application at the Baseline Visit
- Investigational medications or treatments within 30 days of Baseline and during the course of the study

## 5.4 Subject Withdrawal or Removal From Study

As stated in the Informed Consent, all subjects reserve the right to withdraw from the study at any time. An effort will be made to determine why a subject discontinues the study prematurely. The reason for study discontinuation will be recorded in the eCRF. All subjects who terminate the study early and have completed the Baseline Visit will be encouraged to complete Week 26/Early Termination study procedures.

Apr. 23, 2018

Any subject found to have entered the study in violation of this protocol may be withdrawn from the study after discussion with the sponsor. Any subject who requires the use of an unacceptable concomitant medication may be withdrawn from the study. The investigator will discontinue any subject from the study if, in the investigator's opinion, it is not in the subject's best interest to continue.

If the reason for withdrawal is an AE/ SAE, the specific event will be recorded and every effort will be made by the Investigator to document the outcome. The date that the subject is withdrawn from the study and the reason for discontinuation will be recorded on the Case Report Form. Subjects who discontinue from the study or who are lost to follow up will not be replaced.

## 5.4.1 Subject Unblinding Procedures

Randomization lists will be maintained by the sponsor. In case of serious adverse events or other medical emergencies that make it necessary to unblind the treatment code for a specific subject, the investigator will, after consultation with the sponsor, submit a written request for unblinding to the Medical Monitor. The request will be documented, and the applicable information will be sent to the investigator via fax or e-mail. Unblinded subjects will be discontinued from the study.

#### 6 STUDY PROCEDURES

## 6.1.1 Baseline (Qualifying) Visit

Prior to participating in any aspect of the study, each subject will be fully informed, both verbally and in writing, of the conduct and consequences of the study. Each subject must sign the written Informed Consent prior to the conduct of the Baseline (Qualifying) evaluation.

The investigator will assign a unique identification code to each subject being evaluated for participation in the trial. The following procedures will be conducted:


- using the rating guide provided in Appendix A, record right and left Investigator's Global Assessment score of Crow's Feet, both, "at rest" and "on contraction"
- using the same rating guide provided in Appendix A, record right and left Subject's Self-Assessment score of Crow's Feet, both, "at rest" and "on contraction"
- record medical history and concomitant diseases
- record concomitant medication usage
- record history of botulinum use
- female subjects of child-bearing potential will be given a urine pregnancy test
- assess eligibility according to the Inclusion and Exclusion criteria in 5.1 and 5.2

If the subject is deemed eligible to participate in the study, the subject will be randomized and treated.

- record vital signs (weight, height, temperature, resting pulse and blood pressure, and respiration rate)
- collect non-fasting blood samples for laboratory safety testing
- record and transmit a 12-lead ECG
- take color photographs (see Appendix C for photograph procedure)
- evaluate for muscle weakness (ocular and the extremities) or difficulty swallowing or breathing (Signs of Botulinum Toxin Spread, Appendix B)
- provide the study medication with the lowest available Kit No. to the investigator.
- Investigator will apply the topical treatment to the left and right lateral canthal areas
- record subject's experience with the application process
- evaluate for topical adverse event reactions 30 minutes after application using the Irritation Score in Appendix D
- instruct the subject to avoid sun exposure or tanning beds for two days after treatment
- instruct the subject to avoid strenuous activities on the day of application which will cause them to perspire
- instruct the participant not to touch or let others touch the treatment area until the treatment area is washed with soap and water
- instruct the participant to wash the treatment areas with soap and water no sooner than 12 hours after treatment application but no later than 24 hours after treatment application
- schedule follow-up appointment for the next office visit

## 6.1.2 Week 1 Visit (+/- 2 days)

The Week 1 visit will occur one week post Baseline (+/- 2 days):

- ask the open ended "How Do You Feel" question and document answer in the electronic Case Report Form
- if the subject noted any change in well-being since last investigator contact, document details on the Adverse Event eCRF
- record changes in medication usage from the Baseline (Qualifying) visit
- record vital signs (weight, temperature, resting pulse and blood pressure, and respiration rate)
- ask if the subject experienced weakness, lethargy, or difficulty swallowing or breathing
- evaluate for muscle weakness (ocular and the extremities) or difficulty swallowing or breathing (Appendix B)
- using the rating guide provided in Appendix A, record right and left Investigator's Global Assessment score of Crow's Feet, both, "at rest" and "on contraction"
- using the same rating guide provided in Appendix A, record right and left Subject's Self-Assessment score of Crow's Feet, both, "at rest" and "on contraction"
- take color photographs (see Appendix C for photograph procedure)
- schedule the subject for the next office visit

#### 6.1.3 Week 2 Visit (+/- 3 days)

The Week 2 visit will occur two weeks post Baseline (+/- 3 days).

- ask a non-leading "How Do You Feel" question and document answer in the electronic Case Report Form
- if subject noted any change in well-being since last investigator contact, document details on the Adverse Event eCRF
- record changes in medication usage
- record vital signs (weight, temperature, resting pulse and blood pressure, and respiration rate)
- ask if the subject experienced weakness, lethargy, or difficulty swallowing or breathing
- evaluate for muscle weakness (ocular and the extremities) or difficulty swallowing or breathing (Appendix B)
- record and transmit a 12-lead ECG
- using the rating guide provided in Appendix A, record right and left Investigator's Global Assessment score of Crow's Feet, both, "at rest" and "on contraction"
- using the same rating guide provided in Appendix A, record right and left Subject's Self-Assessment score of Crow's Feet, both, "at rest" and "on contraction"

- take color photographs (see Appendix C for photograph procedure)
- schedule subject for the next office visit

## 6.1.4 Week 4 Visit (+/- 4 days)

The Week 4 visit will occur 4 weeks post Baseline +/- 4 days.

- ask a non-leading "How Do You Feel" question and document answer in the electronic Case Report Form
- if subject noted any change in well-being since last investigator contact, document details on the Adverse Event Form
- · record changes in medication usage
- record vital signs (weight, temperature, resting pulse and blood pressure, and respiration rate)
- ask if the subject experienced weakness, lethargy, or difficulty swallowing or breathing
- evaluate for muscle weakness (ocular and the extremities) or difficulty swallowing or breathing (Appendix B)
- using the rating guide provided in Appendix A, record right and left Investigator's Global Assessment score of Crow's Feet, both, "at rest" and "on contraction"
- using the same rating guide provided in Appendix A, record right and left Subject's Self-Assessment score of Crow's Feet, both, "at rest" and "on contraction"
- take color photographs (see Appendix C for photograph procedure)
- · collect non-fasting blood samples for laboratory safety testing
- female subjects of child-bearing potential will be given a urine pregnancy test
- · schedule subject for the next office visit

## 6.1.5 Week 8 Visit (+/- 7 days)

The Week 8 visit will occur 8 weeks post Baseline +/- 7 days.

- ask a non-leading "How Do You Feel" question and document answer in the electronic Case Report Form
- if subject noted any change in well-being since last investigator contact, document details on the Adverse Event Form
- record changes in medication usage
- record vital signs (weight, temperature, resting pulse and blood pressure, and respiration rate)
- using the rating guide provided in Appendix A, record right and left Investigator's Global Assessment score of Crow's Feet, both, "at rest" and "on contraction"
- using the same rating guide provided in Appendix A, record right and left Subject's Self-Assessment score of Crow's Feet, both, "at rest" and "on contraction"
- take color photographs (see Appendix C for photograph procedure)

schedule subject for the next office visit

## 6.1.6 Week 12 Visit (+/- 7 days)

The Week 12 visit will occur 12 weeks post Baseline +/- 7 days.

- ask a non-leading "How Do You Feel" question and document answer in the electronic Case Report Form
- if subject noted any change in well-being since last investigator contact, document details on the Adverse Event Form
- record changes in medication usage
- record vital signs (weight, temperature, resting pulse and blood pressure, and respiration rate)
- using the rating guide provided in Appendix A, record right and left Investigator's Global Assessment score of Crow's Feet, both, "at rest" and "on contraction"
- using the same rating guide provided in Appendix A, record right and left Subject's Self-Assessment score of Crow's Feet, both, "at rest" and "on contraction"
- take color photographs (see Appendix C for photograph procedure)
- schedule subject for the next office visit

## 6.1.7 Week 18 Visit (+/- 7 days)

The Week 18 visit will occur 18 weeks post Baseline +/- 7 days.

- ask a non-leading "How Do You Feel" question and document answer in the electronic Case Report Form
- if subject noted any change in well-being since last investigator contact, document details on the Adverse Event Form
- record changes in medication usage
- record vital signs (weight, temperature, resting pulse and blood pressure, and respiration rate)
- using the rating guide provided in Appendix A, record right and left Investigator's Global Assessment score of Crow's Feet, both, "at rest" and "on contraction"
- using the same rating guide provided in Appendix A, record right and left Subject's Self-Assessment score of Crow's Feet, both, "at rest" and "on contraction"
- take color photographs (see Appendix C for photograph procedure)
- schedule subject for the next office visit

#### 6.1.8 Week 26 Visit (+/- 7 days)

The Week 26 visit will occur 26 weeks post Baseline +/- 7 days.

 ask a non-leading "How Do You Feel" question and document answer in the Case Report Form  if subject noted any change in well-being since last investigator contact, document details on the Adverse Event Form

Apr. 23, 2018

- record changes in medication usage
- record vital signs (weight, temperature, resting pulse and blood pressure, and respiration rate)
- using the rating guide provided in Appendix A, record right and left Investigator's Global Assessment score of Crow's Feet, both, "at rest" and "on contraction"
- using the same rating guide provided in Appendix A, record right and left Subject's Self-Assessment score of Crow's Feet, both, "at rest" and "on contraction"
- take color photographs (see Appendix C for photograph procedure)

## 6.1.9 Study Exit / Early Termination

The scheduled Study Exit is at Week 26. However, if a subject should discontinue prematurely, the following will be performed in addition to the procedures scheduled for the patient's terminating visit:

collect non-fasting blood samples for laboratory safety testing

#### 6.1.10 Unscheduled Visits

The subject may contact the investigator or may be called in for additional unscheduled visits due to safety reasons or at the discretion of the investigator or Sponsor. All unscheduled visits will describe the reason for the visit in the electronic Case Report Form. Some of the procedures that may be completed at an Unscheduled Study Visit are as follows:

- Review of adverse events and concomitant medications
- Vital signs
- Collection of blood samples for laboratory safety testing
- Urine pregnancy testing

#### 7 STUDY DURATION AND CONDUCT

#### 7.1 Conduct of Study

This study will be conducted in compliance with the protocol approved by the Institutional Review Board and according to Good Clinical Practice standards. No intentional deviation from the protocol will be implemented without the prior review and approval of the IRB except where it may be necessary to eliminate an immediate hazard to a research subject. In such case, the deviation will be reported to the IRB as soon as possible.

## 7.2 Duration of Study

Subject enrollment will take approximately 2 weeks per dose group. The total study duration will be approximately 8 months.

Apr. 23, 2018

Each subject will participate for up to 26 weeks. There will be a (Qualifying) Baseline Visit on Week 0 and seven in-office visits at Week 1, 2, 4, 8, 12, 18, and 26.

## 7.3 Stopping Rules

The study is designed as a sequential, overlapping cohort, dose-escalation trial. Enrollment will be halted after each cohort until a safety review has been completed.

- Enrollment into a given cohort and/or proceeding to the next cohort will be halted
  in the event that one serious adverse event (SAE), considered to be probably or
  definitely related to the administration of study medication, is observed.
- Enrollment will be halted in the event that one AE is observed considered to be indicative of distant spread of study medication or unintended exposure to other beings.
- The Sponsor may stop the study in its entirety or discontinue individual study centers at its discretion for any reason or, e.g. if it is observed that the protocol or sound clinical practices are not being followed, or for any other reasons.

The study protocol calls for only one single application of study medication at Baseline (Week 0). Since there is no continuous treatment, no stopping rules for subjects are applicable and subjects will be encouraged to participate in the study until the scheduled termination visit at Week 26.

## 7.4 Monitoring for subject compliance

In this study, a single application of study medication at Day 0 is planned. The study medication will be applied by the Investigator or a designated healthcare professional thereby ensuring compliance with the study application procedure.

Subjects will be queried with regards to concomitant medication at all study visits.

#### 8 ADVERSE EVENT REPORTING

Adverse event reporting will be handled in accordance with the IRB requirements and the requirements of other regulatory authorities that may apply, e.g. the Food and Drug Administration.


Adverse Events reporting will be solicited by non-leading "How Do You Feel" questions. Subtle symptoms of local or systemic spread of toxin effect would be unlikely to be recognized by the subjects as related to treatment. Therefore, study participants will be asked if they experienced weakness, lethargy, or difficulty swallowing or breathing. In addition, information derived from change in concomitant medications, laboratory analyses, and clinical observations will be evaluated for possible indications for side effects. Adverse events resulting from concurrent illnesses or reactions to concurrent medications will also be recorded. The Investigator must monitor the condition of the subject throughout the study from the time of obtaining informed consent until the final study visit.

Any adverse event, including both observed and volunteered problems, complaints, and symptoms, will be recorded on the Adverse Event pages of the electronic Case Report Form. When an adverse event occurs, the following information and assessments should be recorded in the adverse event section of the eCRF:

- The signs, symptoms or diagnosis or the event,
- The date and time of onset of the event using the 24-hour clock where midnight is 00:00 and noon is 12:00. Onset is the date when the first sign or symptoms were first noted.
- Date of recovery/ resolution
- The adverse event severity/ intensity using the criteria outlined in Section 8.1.2
- The relationship of the event to the study drug as outlined in Section 8.1.1
- Any other actions required such as therapy, medication, treatment or diagnostic procedure
- Seriousness of the event using the criteria outlined in Section 8.1.3
- Outcome (recovered, recovered with sequelae, not yet recovered, death)

Follow-up of a subject should be conducted until resolution of the adverse event or until the medical condition is stable. The investigator is responsible for the appropriate medical management of all adverse events.

Adverse events will be analyzed and reported after unblinding of the treatment code within the clinical study report. Serious Adverse Events (SAEs) will be reported by the Sponsor within 10 working days to the IRB as well as the regulatory agency, FDA. In addition, any unanticipated problems involving risk to subjects or others, which in the opinion of the local investigator was unanticipated, serious AND at least possibly related to the research procedures will be reported by the Sponsor to the IRB within 10 working days.

#### 8.1 Definitions

An adverse event is an undesirable or unintentional event affecting the well-being of a subject that occurs during use of the study drug, whether or not considered related to the drug; this includes accidental injuries, reasons for any change in medication (drug and/or dose), and reasons for surgical procedures. It is to be noted that procedures are not adverse events. Abnormal laboratory values or clinically significant changes in laboratory values are not adverse events, but the underlying reasons are. Regardless of the severity or relationship to the investigational drug, all adverse events occurring during the study period must be recorded in the subject's eCRF.

An unexpected adverse event is one that has not been previously observed, or one that is of a specificity or severity not consistent with the current Investigator Brochure.

## 8.1.1 Relationship to Study Drug

The following definitions to assess the causal relationship between an adverse event and the study drug should be used:

Not Related: The event is clearly related to other factors such as a subject's

clinical state, therapeutic interventions or concomitant medications.

Possibly Related: The event has a reasonable temporal relationship to study drug

administration and follows a known response pattern to the study drug. However, a potential alternate etiology may be responsible for

the event.

Related: The event follows a clear-cut temporal sequence from the time of

drug administration and follows a known response pattern to the study drug and either occurs immediately following study drug administration, or improves on stopping the drug, or reappears on

repeat exposure.

#### 8.1.2 Adverse Event Severity

Mild: A mild adverse event is one that the symptoms are barely

noticeable to a subject. It does not influence performance or prevent

a subject from carrying on with normal life activities.

Moderate: A moderate adverse event is one that the symptoms make the

subject uncomfortable and causes some impairment to normal life

activities. Treatment for symptom(s) may be required.

#### Severe:

A severe adverse event is one that the symptoms cause severe discomfort to the subject and severely limits the subject's normal daily activities. Treatment for symptom(s) is given.

Note that "serious" and "severe" are not synonymous. A serious adverse event must fulfill the requirements listed in the definition below, see section 8.1.3.

When intensity changes or occurs more frequently than once a day, the maximum intensity for the event will be listed. If the intensity category changes over a number of days, then these mini-events or changes will be recorded separately (i.e., having distinct onset days).

#### 8.1.3 Serious Adverse Events

A serious adverse event is an event that is:

- fatal / results in death
- life-threatening
- results in persistent or significant disability/incapacity
- requires or prolongs subject hospitalization or
- is a congenital anomaly or birth defect.

<u>Life Threatening</u> is defined as an event in which a subject is at risk of death at the time of the event. It does not refer to an event that hypothetically might have caused death if it was more severe.

<u>Death</u>: The death of an enrolled subject is not an event, but an outcome. It is the event that resulted in a fatal outcome that must be reported.

<u>Disability</u> is defined as a substantial disruption of a person's ability to conduct normal life functions.

ANY SERIOUS ADVERSE EVENT, INCLUDING DEATH DUE TO ANY CAUSE, WHICH OCCURS DURING THIS INVESTIGATION, WHETHER OR NOT RELATED TO THE STUDY MEDICATION, MUST BE REPORTED **IMMEDIATELY** (DURING NORMAL BUSINESS HOURS, 9 AM TO 5 PM, ET) TO THE SPONSOR/MEDICAL MONITOR.

Any serious adverse event should be reported to Eirion Therapeutics by telephone or fax within 24 hours of the event. The call should be followed-up with the completion of the written SAE report form within five days of receiving firsthand knowledge of the event. Full details of the event, any sequelae and an assessment of the relationship to the study drug must be provided in the report. Any serious adverse event must also be reported to the Institutional Review Board within 48 hours of receiving firsthand knowledge of the

event and a copy of this SAE report must be sent to Eirion Therapeutics. The original SAE report form should be maintained in the Regulatory Binder. It is the Sponsor's responsibility to fulfill reporting obligations to the FDA.

Reports of serious adverse events should be made by telephone to:

Eirion Therapeutics Clinical Development Department: 215-356-7532 (phone)

888-664-2736 (fax)

Serious adverse events associated with the use of the study medication will be reported to appropriate regulatory agencies, investigators, and the IRB by the Sponsor.

## 8.1.4 Unanticipated Problems Involving Risk to Subjects or Others

Unanticipated problems involving risk to subjects or others are:

- Any serious event (including on-site and off-site adverse events, injuries, side
  effects, deaths or other problems) which in the opinion of the local investigator was
  unanticipated, involved risk to subjects or others, and was possibly related to the
  research procedures.
- Any serious accidental or unintentional change to the IRB-approved protocol that involves risk or has the potential to recur.
- Any deviation from the protocol taken without prior IRB review to eliminate apparent immediate hazard to a research subject.
- Any breach in confidentiality that may involve risk to the subject or others.
- Any other serious and possibly related event which in the opinion of the investigator constitutes an unanticipated risk.

## 8.2 Adverse Event Follow-up

Adverse events and Serious Adverse Events will be followed up until their resolution or until a stable outcome has emerged.

## 8.2.1 Pregnancy

Every effort must be made to avoid pregnancy during the study. If pregnancy does occur, Eirion Therapeutics must be informed immediately. The mother and fetus must be followed until the birth of the infant. In general, the follow up will include the course, duration, and outcome of the pregnancy, and the infant outcome. As the investigational product is applied only once during the study, subjects having a positive urine pregnancy test at or after the Week 4 Visit will be permitted to remain in the study.

Medically accepted methods of birth control are surgical sterilization (tubal sterilization or hysterectomy), vaginal ring contraceptive, patch contraceptive, injectable contraceptive,

implantable contraceptive, Intrauterine Device (IUD), diaphragm, condom, or spermicidal gel or foam. Oral contraceptives (prescribed birth control pill) are also acceptable provided this method has been used for at least 4 months prior to the qualifying visit with no change of the brand within this period.

#### 9 STATISTICAL PLAN

#### 9.1 Statistical Methods

## 9.1.1 Study Population

Due to the dose sequential study design with each cohort containing both active and placebo-treated subjects, a subset of safety and efficacy analyses (Cohort Analyses) will be performed after each cohort has completed the Week 4 visit on data from the most recent cohort. The full set of safety and efficacy analyses (Final Analysis) will be performed on data from all completed cohorts after all subjects have completed the study. The Final Analysis will treat all Vehicle data across Cohorts as one treatment group. Because of the small number of Vehicle subjects in each Cohort, p-values from Cohort Analyses will be reviewed for general directional guidance only and will not be expected to reach statistical significance. The following sections will apply to both Cohort and Final Analyses if no distinction is made.

Descriptive statistics will be used to summarize demographic characteristics (age, gender, race, height and weight) and background characteristics for all randomized subjects by treatment group. Past/coexistent medical history information for all randomized subjects will be presented in a by-subject listing. Baseline assessments of LCL severity will also be presented as background characteristics of the population and summarized by treatment group.

Demographic data will be summarized using descriptive statistics. Categorical measures will be summarized by counts and percentages. Continuous measures will be summarized with means, standard deviations and ranges (min and max).

Descriptive statistics will be used to summarize study medication compliance and exposure for all randomized subjects. Prior and concomitant medication information for all enrolled subjects will be presented in a by-subject listing.

#### 9.1.2 Primary Efficacy Analysis

Unless otherwise specified, efficacy analyses are based on the findings for the treatment area, i.e. lateral canthal area only. Alpha will be set at 0.05 using two-tailed tests. The Crow's Feet Wrinkle scale is an ordinal categorical variable ranging from 0 to 4. The

investigator's assessment will be summarized for each treatment group and at each visit using frequency distributions. IGA data will be analyzed at Week 4, 8, and Week 12 to evaluate the proportion of patients achieving treatment success, defined as None (0), Minimal (1) or Mild (2), using a Chi-square test. The primary efficacy analysis will be for each cohort separately, and for all cohorts pooled where the Vehicle group will include subjects randomized to vehicle across all cohorts.

Apr. 23, 2018

## 9.1.3 Secondary Efficacy Analyses

As secondary efficacy analysis data will be analyzed at Week 4, 8, and Week 12 to evaluate the proportion of patients achieving a composite treatment success, defined as None, Minimal, or Mild (0 - 2), in both the IGA and the SSA.

In addition, Change from Baseline in the Investigator's Global Assessment Score, will be analyzed using a one-way analysis of variance (ANOVA). Planned pairwise comparisons of each dose group with Vehicle will be made within the ANOVA model using LSMeans and the pooled error term, with no alpha adjustment for multiple comparisons. An analysis of covariance (ANCOVA) with baseline average IGA score as the covariate will be used if it yields greater sensitivity than the ANOVA model.

Secondary end-points will include the average of right and left canthal area IGA score at rest, and the subject self-assessment at rest and on contraction, for overall condition and responder analyses defined as Change From Baseline by 1 or 2 ordinals. Each analysis will use the same statistical methods as described for the Primary Efficacy Analysis. In addition, similar analyses will be performed for each post-baseline visit not covered in the Primary Efficacy Analysis. In the event that a clinically significant number of subjects have different IGA-LCL Scores in right and left canthal areas at Baseline, a similar IGA-LCL Score analysis will be performed on the canthal area for each subject with the greatest score at baseline. The same ANOVA or ANCOVA model as above will be employed to evaluate statistical significance of the overall dose response using an appropriate linear contrast within the model, where Vehicle is treated as a dose of 0.0 U.

#### 9.1.4 Safety Analysis

The assessment of safety will be based mainly on the frequency of adverse events. Other safety data (e.g., vital signs and special tests) will be summarized as appropriate.

Adverse events will be coded using a current MedDRA dictionary and summarized by presenting, for each treatment group, the number and percentage of subjects having any adverse event, having an adverse event in each body system (System Organ Class), and having each coded individual adverse event. Other adverse event information collected (e.g., severity/intensity or relationship to study medication) will be listed as appropriate.

Data from other tests will be listed, notable values will be flagged, and any other information collected will be listed as appropriate. No inferential statistical tests are planned for safety data but may be performed on an ad-hoc basis to highlight any comparisons that may warrant further consideration.

## 9.2 Subject Population(s) for Analysis

## 9.2.1 Sample size

This study is powered based on the results from published studies using similar active ingredients.

## 9.2.2 ITT and PP population

Statistical analysis of efficacy will be performed on the ITT population of all treated subjects with at least one post-baseline visit, including those for whom only incomplete data are available.

Where data are missing due to subject discontinuation or other reasons, the last post-baseline observation carried forward (LOCF) procedure will be used for each post-baseline visit with missing data. Subjects who are lost to follow-up who do not have at least one post-baseline visit will not be included in the analysis.

An additional analysis may be performed in the per protocol population. Subjects will be considered "per protocol" if they complete the Week 26 evaluation without noteworthy protocol violation. No data imputations will be made for this analysis.

## 9.3 Significance

Unless otherwise specified, all statistical tests will be conducted against a two-sided alternative hypothesis, employing a significance level of 0.05.

#### 9.4 Termination Criteria

Enrollment into the study will be halted as described in section 7.3 Stopping Rules. Safety assessments between Cohorts will be used to confirm continuation of the study to the next Cohort. No other type of interim analysis is planned that could trigger termination of the trial

#### 9.5 Deviation Reporting

A Statistical Analysis Plan will be created prior to the completion of the study and unblinding of the database. Any deviations from or additions to the statistical analyses specified in the protocol will be described and justified in the Statistical Analysis Plan.

#### 10 DIRECT ACCESS TO SOURCE DATA/DOCUMENTATION

Data reflecting subject experience with the drug under investigation will be recorded on appropriate source documents and in the eCRF. The investigator understands that the office and hospital records of subjects entered in this study will be required to be available to copying and inspection if requested by a properly authorized employee of the Sponsor or the Department of Health and Human Services, under the supervision of the investigator or a designated representative and in accordance with Federal regulations.

#### 11 QUALITY CONTROL AND QUALITY ASSURANCE

The investigator will allow Eirion Therapeutics or their designated affiliates to periodically audit, at mutually convenient times during the study and after the study has been completed, all source documents and corresponding portions of office, hospital, and laboratory records of each subject. The monitoring visits will provide Eirion Therapeutics with the opportunity to confirm the rights and safety of the subjects, ensure the confidentiality of the data and subject's identification, evaluate the progress of the study, verify the accuracy and completeness of the eCRFs, assure compliance with protocol requirements, applicable FDA regulations, IRB and ICH-GCP Guidelines, confirm that investigator's obligations are being fulfilled, and resolve any inconsistencies in the study records. The sponsor may stop the study if it is observed that the protocol or sound clinical practices are not being followed.

## 12 ETHICAL CONSIDERATIONS

This study must be approved by an IRB or other ethical approval body prior to subject enrollment. The governing IRB must comply with all the requirements set forth in 21 CFR § 56. The IRB is responsible for the initial approval, any amendments, advertisements, and continuing review of the proposed clinical study. The IRB will review any written materials given to the subject and the Informed Consent Forms. The investigator must retain a copy of the approval letter that contains the study number, protocol title and identification of all documents approved. A copy of the letter must be sent to the sponsor prior to drug shipment to the investigator.

The investigator agrees to promptly report to the IRB all unanticipated problems involving risks to human subjects or others.

The investigator will ensure that this study is conducted in full conformity with the principles of the "Declaration of Helsinki" and with the laws and regulations of the participating countries, whichever affords the greater protection to the individual. It is the responsibility of the investigator to obtain informed consent in written form (according to

local legal requirements) from each subject participating in this study. All subjects will be informed of the aims, methods, anticipated benefits, potential hazards and confidentiality of data. Candidates will also be told that they are free to refuse participation or withdraw from the study at any time. A consent form must be signed and dated by the subject before he/ she is exposed to any study-related procedure, including screening tests for eligibility. The subject will receive a copy of the signed consent. The subject should be informed if new information becomes available that may be relevant to his/ her willingness to continue participation in the study. Each subject will be informed that the monitor, in accordance with applicable regulatory requirements, may review his/ her medical records and data.

Periodic status reports must be submitted at least yearly to the IRB. Within three months after completion or termination of the study, a final report should be submitted to the IRB and the Sponsor. The investigator must maintain an accurate and complete record of all submissions made to the IRB including a list of all reports and documents submitted.

The investigator is responsible for maintaining all the records which enable the conduct of the study at the site to be fully understood in compliance with the ICH-GCP filing standard. The investigator is responsible for the completion and maintenance of the confidential subject identification code which provides the sole link between named subject source records and the eCRF data. The investigator must arrange for the retention of study records for 5 years after the completion of the study. No study site files may be destroyed without prior written agreement between the investigator and the sponsor. Should the investigator elect to assign the study documents to another party, or move them to another location not noted on the FDA 1572 Form, the sponsor must be notified.

#### 13 DATA HANDLING AND RECORD KEEPING

Data reflecting subject experience with the drug under investigation will be recorded in the eCRF. Sites may use a print-out of the eCRF or their own record keeping system as source documentation. After monitoring, source verification and authentication by the Principal Investigator, the eCRF will be locked. The study specific data in the eCRF are the sole property of the Sponsor.

It is the Investigator's responsibility to ensure completion and to review and approve all data in the eCRF and source documents. At all times, the Investigator has final responsibility for the accuracy and authenticity of all clinical and laboratory data entered on the eCRF and source document.

All fields and blanks must be completed or marked intentionally blank as appropriate following the instructions on the eCRF. eCRFs will be electronically signed and dated by the investigator or a designated representative. If an entry on an eCRF already submitted requires change, the Electronic Data Capture (EDC) system will capture the reason for the change and then the correction will be made according to the procedures dictated by the EDC system.

The investigator will maintain adequate records for the study including subject's eCRFs, medical records, laboratory reports, informed consent forms, drug accountability records, safety reports, information regarding subjects who discontinued, and any other pertinent data.

#### 14 FINANCE

The study will be sponsored by Eirion Therapeutics, Inc.

#### 15 INVESTIGATOR'S AGREEMENT

I have read Eirion Therapeutics' protocol entitled: "Clinical Trial to Evaluate ET-01 in Subjects with Lateral Canthal Lines" in conjunction with the "Investigators Drug Brochure" which contains all information necessary to the conduct of the study. I agree to conduct the study as outlined therein and according to ICH Good Clinical Practice.

Investigator's Signature Date

Apr. 23, 2018

Sponsor's Signature Date

Klaus Theobald, MD, PhD
Chief R&D Officer
Eirion Therapeutics, Inc.

#### 16 REFERENCES

Ascher, Benjamin; Rzany, Berthold; Grover, Rajiv Efficacy and Safety of Botulinum Toxin Type A in the Treatment of Lateral Crow's Feet: Double-Blind, Placebo-Controlled, Dose-Ranging Study Dermatol Surg 35:1478-1486, 2009

Carruthers, Alastair; Carruthers, Jean; Hardas, Bhushan; Kaur, Mandeep; Goertelmeyer, Roman; Jones, Derek; Rzany, Berthold; Cohen, Joel; Kerscher, Martina; Corcoran Flynn, Timothy; Maas, Corey; Sattler, Gerhard; Gebauer, Alexander; Pooth, Rainer; McClure, Kathleen; Simone-Korbel, Ulli; Buchner, Larry A Validated Grading Scale for Crow's Feet Dermatol Surg 2008; 34:S173–S178

Coté, Timothy; Mohan, Aparna; Polder, Jacquelyn; Walton, Marc; Braun, Miles Botulinum toxin type A injections: Adverse events reported to the US Food and Drug Administration in therapeutic and cosmetic cases
J. Am. Acad. Dermatol. 2005;53:407-15

# **Appendix A: Crow's Feet Wrinkle Scale1**

The Crow's Feet Wrinkle Scale (CFW) is a photonumeric guide that grades severity of lateral canthal lines according to one of the following five descriptions.

| Score | Grade | Description | At Rest | At Smile |
|---|---|---|---|---|
| 0 | Absent | No visible wrinkles | | |
| 1 | Minimal | Very fine wrinkles (that are barely visible) | | |
| 2 | Mild | Fine wrinkles (that are shallow) | | |
| 3 | Moderat<br>e | Moderate wrinkles (that are moderately deep) | | |
| 4 | Severe | Severe wrinkles (that are severely deep) | | |

<sup>1</sup> Carruthers et. al. A Validated Grading Scale for Crow's Feet, Dermatol Surg 2008; 34:S173–S178

Confidential

Investigators and subjects will use the same scale. As a photo guide, the guidance pictures shown below will be presented as 11" x 17" laminated poster cards.

Instructions for use:

## For Investigators:

- "At Rest": Ask the subject to make an expressionless face and indicate with a check mark the description that best describes his/her appearance.
- "On Contraction": Ask the subject to make a maximally exaggerated smile and indicate with a check mark the description that best describes his/her appearance.

## For Subjects:

- Place the subject in front of a mirror or provide a hand-held mirror in a well lit room
- Provide subject with the photo guide
- "At Rest": Ask the subject to make an expressionless face and state the grade that best describes his/her appearance. Record in the eCRF.
- "On Contraction": Ask the subject to make a maximally exaggerated smile and using the provided scale state the grade that best describes his/her appearance.
   Record in the eCRF.

# **Appendix B: Signs of Botulinum Toxin Spread**

- 1. Ask the subject to follow the examiner's finger with his or her eyes without moving his or her head. At eye level, the examiner should move his or her finger to the right of the subject's head and then to the left. Repeat this horizontal motion at the level of the subject's forehead and chin. Note whether there is any abnormality in the form of any inability of the subject's eyes to follow the finger.
- 2. Ask the subject to raise his/her eyelids. Observe any indication for "drooping".
- 3. Ask the subject to swallow and note any difficulty doing so.
- 4. Ask the subject to partially flex his or her arms at the elbow, with fist at shoulder level. Ask the subject to attempt to fully flex his or her arms against the resistance of the examiner pulling on the subject's forearms. Note whether there is an abnormality in the form of any muscular weakness.
- 5. Ask the subject to squat down and stand up again. Watch for any abnormalities or signs of weakness.

# **Appendix C: Procedure for Color Photography**

Equipment: Digital Camera, Log Book, Subject-Specific Index Card

Procedure:

In these clinical photographs, for the duration of the study, the only variable allowed to change is the skin condition itself. Therefore, anything extraneous to the condition (jewelry, makeup, clothing, furniture, walls, etc.) is to be eliminated from the fields to be photographed, from baseline through the final photographs. The necessity of good photos should be stressed to the subjects to ensure their cooperation. Camera, lighting, framing, and exposure must be held consistent. In the end, the pictures should read like a time-lapse movie.

Ask the subject to stand against a light background, away from any window or other source of external light. The subject should hold a white index card with his/her identification number and initials. The photographer should stand about 1 foot away from the subject and set the camera for minimum zoom and take 5 photographs: 1 full frontal face photo, and one 45° view of each of the right and left periorbital region, both, "at rest" and "on contraction".

For the "at rest" pictures, ask the subject to have a relaxed, expressionless composure. In the frontal picture, the subject should hold an index card with subject ID, date and initials. The ID card is not required for the 45° views. For the "on contraction" pictures, ask the subject to produce a smile that is maximally exaggerated by exhorting the subject to make the biggest smile possible.

Maintain a Log Book that includes the following information:

- Protocol Number
- Investigator Name
- Subject Initials
- Subject ID Number
- Visit week
- Date of Visit
- Photographer's Initials

At monitoring visits, the Study Monitor will upload the pictures from the camera to a laptop computer.

# **Appendix D: Irritation Scoring**

For the irritation assessment, the following scale will be utilized:

#### Numeric Grades:

- 0 = no evidence of irritation
- 1 = minimal erythema, barely perceptible
- 2 = definite erythema, readily visible; or minimal edema; or minimal papular response
- 3 = erythema and papules
- 4 = definite edema
- 5 = erythema, edema, and papules
- 6 = vesicular eruption
- 7 = strong reaction spreading beyond test site

All clinically significant skin responses observed with the test products or any score of 3 or higher will be reported as an adverse event.